CLINICAL TRIAL: NCT04293172
Title: A Randomised, Double Blind, Parallel Group, Multicentre, Phase III Study to Evaluate the Effect of Ticagrelor Versus Placebo in Reducing the Number of Vaso-Occlusive Crises in Paediatric Patients Aged 6 Months to <18 Years With Sickle Cell Disease (HESTIA5)
Brief Title: Study to Evaluate the Effect of Ticagrelor Versus Placebo in Reducing Vaso-Occlusive Crises Rate in Pediatric Patients With Sickle Cell Disease.
Acronym: HESTIA5
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrolment of first patient.
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5136C00013
Record Dates: First submitted 2020-02-04; First posted 2020-03-03 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Disease
Keywords: Ticagrelor; Vaso-Occlusive Crises; Paediatric Patients; 6 Months to <18 Years; Sickle Cell Disease; Sickle Cell Anemia; Platelet aggregation; Brillinta; Acute Chest Syndrome; painful crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Experimental): The double-blinded study drug dose will be weight dependent.
  Interventions: Drug: Brilinta
- Placebo (Placebo Comparator): The double-blinded study drug dose will be weight dependent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brilinta — Patients in the open-label Run-in period (patients aged 6 to <24 months only) will receive ticagrelor 5 mg twice a day (body weight 6 to ≤9 kg), 10 mg twice a day (body weight >9 to ≤12 kg) or 15 mg twice a day (body weight >12 to ≤24 kg) for 14 days.
  The double-blind IP will be based on 5 weight bands:
  * 6 to ≤9 kg: ticagrelor 5 mg or matching placebo, twice a day
  * >9 to ≤12 kg: ticagrelor 10 mg or matching placebo, twice a day
  * >12 to ≤24 kg: ticagrelor 15 mg or matching placebo, twice a day
  * >24 to ≤48 kg: ticagrelor 30 mg or matching placebo, twice a day
  * >48 kg: ticagrelor 45 mg or matching placebo, twice a day
  Arms: Ticagrelor
Drug: Placebo — Patients in the open-label Run-in period (patients aged 6 to <24 months only) will receive ticagrelor 5 mg twice a day (body weight 6 to ≤9 kg), 10 mg twice a day (body weight >9 to ≤12 kg) or 15 mg twice a day (body weight >12 to ≤24 kg) for 14 days.
  The double-blind IP will be based on 5 weight bands:
  * 6 to ≤9 kg: ticagrelor 5 mg or matching placebo, twice a day
  * >9 to ≤12 kg: ticagrelor 10 mg or matching placebo, twice a day
  * >12 to ≤24 kg: ticagrelor 15 mg or matching placebo, twice a day
  * >24 to ≤48 kg: ticagrelor 30 mg or matching placebo, twice a day
  * >48 kg: ticagrelor 45 mg or matching placebo, twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of ticagrelor vs placebo for the reduction of Vaso-Occlusive crises in paediatric patients with Sickle Cell Disease

DETAILED DESCRIPTION:
* HESTIA5 will evaluate the efficacy, safety and tolerability of ticagrelor versus placebo in children with SICKLE CELL DISEASE during treatment for at least 12 months and up to a maximum of 24 months.
* The target population are children (males and females) aged 6 months to <18 years and body weight ≥6 kg diagnosed with homozygous sickle cell or sickle beta-zero-thalassaemia confirmed by high-performance liquid chromatography or hemoglobin electrophoresis. The aim is to randomise 20 patients in the age group 6 to <24 months. At least 50 patients should be randomised in each of the age groups: ≥2 to <12 years and ≥12 to <18 years.
* Prior to randomisation in this study, patients aged 6 to <24 months will undergo a 14-day Run in period in which they will receive open-label ticagrelor twice a day for 14 days according to weight. Run-in period includes 4 visits, called R1, R2, R3 and R4. The run-In period is to ensure that the treatment is well-tolerated, and that the exposure is in line with model-based predictions following repeated twice a day dosing with ticagrelor in this age group. At the end of the Run-in period (Visit R4), the patient will take his/her final dose of open-label IP and await the independent Data Monitoring Committee chairman's evaluation of tolerability, safety and exposure before being eligible to enter the Screening period for randomisation. Patients who complete the Run-in period according to the protocol must also meet all the inclusion/exclusion criteria detailed in Protocol, to proceed to randomisation.
* To be eligible for the study, patients must have experienced at least 2 VASO-OCCLUSIVE CRISES (defined as painful crisis and/or ACUTE CHEST SYNDROME) events in the past 12 months prior to Visit 1, (patients aged 2 to <18 years) and prior to visit R1 (patients aged 6 to <24 months) indicating that the severity of the patient's disease justifies preventive chronic long-term treatment. Even if painful VASO-OCCLUSIVE CRISES are uncommon in infants and become more frequent in older children, data show that symptoms like dactylitis precede more severe events and confirm that children who have early dactylitis are more likely to have severe events later in life.
* Study participants should receive standard of care for SICKLE CELL DISEASE, adjusted to the individual patient at the discretion of the investigator, including routine health care screening examinations and immunizations to local guidelines and health care programmes. Study drug will be given on the background of standard treatments for SICKLE CELL DISEASE. Study participants are not withheld from any other treatments that may be used in SICKLE CELL DISEASE (eg., hydroxyurea) during the trial, which is important considering the use of a placebo control group. However, restrictions apply to some medications and interventions that may be necessary for the patient's health and well-being during the study.
* Patients are to be followed until a common study end date (CSED) is reached defined as 12 months after the last patient is randomized. Treatment duration is at least 12 months for study participants, and patients will continue on treatment until 12 months after last randomized patient or up to a maximum of 24 months. The expected average follow-up is 18 months, assuming a uniformly distributed enrolment period of 12 months. Considering inclusion of patients with at least 2 VASO-OCCLUSIVE CRISES in the past year, this treatment duration is considered long enough to evaluate effects on VASO-OCCLUSIVE CRISES events as well as to capture safety and tolerability data supporting a potential future long term use of ticagrelor.
* Due to ticagrelor mechanism of action and the potential to reduce symptoms caused by ischemia during a vaso-occlusion, a composite endpoint with painful crises and/or ACUTE CHEST SYNDROME has been selected for the primary endpoint. Painful crisis is the most common reason for emergency department visits for patients with SICKLE CELL DISEASE with a significant impact on young patients' lives, affecting them physically and emotionally. Secondary endpoints are included to broaden the understanding of effects in patients with SICKLE CELL DISEASE and to also assess potential benefits on symptomatic disease burden and health-related quality of life (HRQL).
* Patients will be treated with 5, 10, 15, 30 and 45 mg twice a day or matching placebo, depending on body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures not part of standard medical care (local regulations and international guidelines are to be followed in determining the assent/consent requirements for children).
2. Children aged 6 months to <18 years of age and body weight ≥6 kg diagnosed with HbSS or HbS/β0 as confirmed by high-performance liquid chromatography (HPLC) or haemoglobin electrophoresis.
3. Have experienced at least 2 VASO-OCCLUSIVE CRISES (painful crisis and/or ACUTE CHEST SYNDROME) as judged by the Investigator in the past 12 months prior to Visit R1 (patients aged 6 to <24 months) or Visit 1 (patients aged 2 to <18 years). These VASO-OCCLUSIVE CRISES need to be documented in the patient's medical records or in other documents that can be reconciled.
4. If aged 2 to ≤16 years, must have had a TCD within the past year prior to Visit 2. If this is not the case, a TCD examination must be done before randomisation.
5. If aged ≥10 years, must have had an ophthalmological examination within the past year prior to Visit 1. If this is not the case, the patient must be examined by an ophthalmologist before proceeding in the study. If local guidelines dictate ophthalmological examination at younger ages, those local guidelines should be followed.
6. If treated with hydroxyurea or L-glutamine, the weight-adjusted dose must be stable for 3 months before screening.
7. Suitable venous access for the study-related blood sampling.
8. Prior to dosing on day of randomisation (Visit 2), a negative urine (dipstick) pregnancy test performed at Enrolment (Visit 1) and at Visit 2 must be available for female patients of childbearing potential.
9. Females of childbearing potential (after menarche) must not become pregnant during the study. Sexually active females must use a highly effective method of contraception which results in a low failure rate (ie, less than 1% per year). If use of effective contraception cannot be secured in sexually active females, the patient cannot be included in this study.

Exclusion Criteria:

1. As judged by the Investigator, any evidence of unsuitability which in the Investigator's opinion makes it undesirable for the patient to participate in the study.
2. History of transient ischaemic attack (TIA) or cerebrovascular accident (ischaemic or haemorrhagic), severe head trauma, intracranial haemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy.
3. Findings on TCD: Current or previous values for time averaged mean of the maximum velocity (TAMMV) that are Conditional or Abnormal. Patients with Conditional TAMMV values or higher (≥153 cm/sec using TCD imaging technique [TCDi] which is corresponding to ≥170 cm/sec by the non-imaging technique). Both the middle cerebral artery and the internal carotid artery should be considered. Any other criteria that would locally be considered as TCD indications for chronic transfusion would also exclude the patient.
4. Pathological finding on any other imaging assay indicating increased risk for intracerebral bleeding or thromboembolism.
5. International normalised ratio (INR) >1.4 or active pathological bleeding or increased risk of bleeding complications according to Investigator.
6. Haemoglobin <6 g/dL from test performed at Visit R1 and Visit 1 (patients aged 6 to <24 months) or at Enrolment (Visit 1) (patients aged 2 to <18 years).
7. Platelets <100 × 109/L from test performed at Visit R1 and Visit 1 (patients aged 6 to <24 months) or at Enrolment (Visit 1) (patients aged 2 to <18 years).
8. Undergoing treatment with chronic red blood cell transfusion therapy.
9. Chronic use of NSAIDs defined as continuous intake >3 days per week that cannot be discontinued.
10. Receiving chronic treatment with anticoagulants or antiplatelet drugs that cannot be discontinued.
11. Moderate or severe hepatic impairment defined as laboratory values of alanine aminotransferase (ALT) >2×upper limit of normal (ULN), total bilirubin >2×ULN (unless judged by the Investigator to be caused by haemolysis), albumin <35 g/L (3.5 g/dL) and INR >1.4, or symptoms of liver disease (eg, ascites) from test performed at Visit R1 and Visit 1 (patients aged 6 to <24 months) or at Enrolment (Visit 1) (patients aged 2 to <18 years).
12. Renal failure requiring dialysis.
13. Patient considered to be at risk of bradycardic events (eg, known sick sinus syndrome or second- or third-degree atrioventricular block) unless already treated with a permanent pacemaker.
14. Concomitant oral or intravenous therapy with strong cytochrome P450 3A (CYP3A) inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers, which cannot be stopped at least 5 half-lives before randomisation.
15. Active untreated malaria. Patients with suspected malaria at Visit R1 (patients aged 6 to <24 months) or at Enrolment (Visit 1) (patients aged 2 to <18 years) will be tested.
16. Known hypersensitivity or contraindication to ticagrelor.
17. Patients who are currently pregnant or breastfeeding or planning to become pregnant during the study or have given birth less than 3 months prior to Enrolment (Visit 1).
18. Concern for the inability of the patient or caregiver (defined as legally authorised representative) to comply with study procedures and/or follow-up.
19. Previous randomisation in the present study or participation in any previous HESTIA study.
20. Participation in another clinical study with an IP or device during the last 30 days preceding screening.
21. Involvement of member of patient's family, or patient self, in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of Vaso-Occlusive Crises | Up to end of study visit (12 to 24 months)
  Vaso-occlusive crises (VOC) defined as the composite of a painful crisis and/or an Acute Chest Syndrome (ACS) . Each component is defined as:
  A painful crisis is an onset or worsening of pain that lasts at least 2 hours, for which there is no explanation other than vaso-occlusion and which requires therapy with oral or parenteral opioids, parenteral NSAIDs, or other analgesics prescribed by a health care provider in a medical setting (such as a hospital, clinic or emergency room visit) or at home.
  An ACS is an acute illness characterized by fever and/or respiratory symptoms, accompanied by a new pulmonary infiltrate on a chest X-ray.

SECONDARY OUTCOMES:
Number of Vaso-Occlusive Crises in patients aged 2 to <18 years | Up to end of study visit (12 to 24 months)
Number of painful crises | Up to end of study visit (12 to 24 months)
Number of Acute Chest Syndromes | Up to end of study visit (12 to 24 months)
Duration of painful crises | Up to end of study visit (12 to 24 months)
Number of Vaso-Occlusive Crises requiring hospitalisation or emergency department visits | Up to end of study visit (12 to 24 months)
Number of days hospitalised for Vaso-Occlusive Crises | Up to end of study visit (12 to 24 months)
Number of acute Sickle Cell Disease complications | Up to end of study visit (12 to 24 months)
Number of days hospitalised for acute Sickle Cell Disease complications | Up to end of study visit (12 to 24 months)
Number of sickle cell-related red blood cell (RBC) transfusions | Up to end of study visit (12 to 24 months)
Health-related quality of life (HRQL) | At randomization, visit 9 (6 months), visit 15 (12 months), visit 21 (18 months) and End of Study visit (12 to 24 months).
  HRQL total score and by dimension using Paediatric Quality of Life Inventory (PedsQL) Sickle Cell Disease Module; and Fatigue total score and by dimension using the PedsQL Multidimensional Fatigue Scale (age appropriate versions: 2 to 4 years; 5 to 7 years; 8 to 12 years; 13 to 18 years); HRQL total score and by dimension using the PedsQL Infant Scale (age appropriate versions: 1 to 12 months; 13 to 24 months)
Absence from school or work due to Sickle Cell Disease | Up to end of study visit (12 to 24 months)
  Proportion of days of absence from school or work (only if going to school or work at randomisation)
Intensity of pain during Vaso-Occlusive Crises in patients aged ≤4 years | Up to end of study visit (12 to 24 months)
  Intensity of worst pain daily during Vaso-Occlusive Crises
  - For patients aged ≤4 years, observer reported using the Face, Legs, Activity, Cry, Consolability (FLACC) scale
Intensity of pain during Vaso-Occlusive Crises for patients aged 5 to <18 years | Up to end of study visit (12 to 24 months)
  Intensity of worst pain daily during Vaso-Occlusive Crises
  - For patients aged 5 to <18 years, self-reported using the Faces Pain Scale - Revised (FPS-R)
Type of analgesics (opioid and non-opioid) use | Up to end of study visit (12 to 24 months)
Palatability and Swallowability | Immediately after administration of IP at randomization and visit 9 (6 months)
  For patients aged ≤4 years taking the tablet dispersed or whole, an observer assessment of palatability will be undertaken
Palatability and Swallowabilty | Immediately after administration of IP at randomization and visit 9 (6 months)
  For patients aged ≥5 years taking the tablet dispersed or whole, palatability will be assessed and categorised using the Facial Hedonic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Anders Berggren, MD, PhD, Study Director — AstraZeneca